CLINICAL TRIAL: NCT00902330
Title: Cranial Stimulation for Chemotherapy Symptoms in Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: MCC-11995; HM11995 (Other: VCU IRB); CDR0000641994 (Registry Identifier: PDQ (Physician Data Query)); NCI-2011-00234 (Registry Identifier: CTRP (Clinical Trials Reporting System))
Record Dates: First submitted 2009-05-14; First posted 2009-05-15 (Estimated); Results first posted 2015-04-02 (Estimated); Last update posted 2015-11-23 (Estimated); Status verified 2015-11

CONDITIONS: Anxiety Disorder; Breast Cancer; Depression; Fatigue; Pain; Sleep Disorders
Keywords: depression; anxiety disorder; fatigue; pain; sleep disorders; stage IA breast cancer; stage IB breast cancer; stage II breast cancer; stage IIIA breast cancer
MeSH Terms: conditions — Anxiety Disorders; Breast Neoplasms; Depression; Fatigue; Pain; Sleep Wake Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (cranial microcurrent electrical stimulation [CES]) (Experimental): Patients receive a CES unit (Alpha-Stim® 100 Microcurrent Stimulator) that passes microcurrent levels of biphasic electrical stimulation via ear-lobe electrodes. The CES unit is preset to provide 1 hour of 100 μA (sub-sensory level), modified square-wave biphasic stimulation on a 50% duty cycle at .05 Hz, and to automatically turn off at the end of 1 hour. Patients use their CES unit once daily in weeks 1-18.
  Interventions: Procedure: energy-based therapy
- Arm II (sham CES) (Sham Comparator): Patients receive a CES unit as in arm I, but the ear-lobe electrodes do not pass electrical current. Patients use their CES unit once daily in weeks 1-18.
  Interventions: Procedure: sham intervention

INTERVENTIONS:
Procedure: energy-based therapy — Given once a day for 18 weeks
  Arms: Arm I (cranial microcurrent electrical stimulation [CES])
Procedure: sham intervention — Given once a day for 18 weeks
  Arms: Arm II (sham CES)

SUMMARY:
RATIONALE: Cranial microcurrent electrical stimulation (CES) is mild electrical current received through electrodes placed on the earlobes. CES may lessen symptoms in women with breast cancer receiving chemotherapy. It is not yet known whether CES is more effective than sham therapy in reducing symptoms caused by chemotherapy in women with breast cancer.

PURPOSE: This randomized phase III trial is studying mild electrical stimulation to see how well it works compared with sham therapy in reducing symptoms caused by chemotherapy in women with stage I, stage II, or stage IIIA breast cancer receiving chemotherapy.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To compare the effects of cranial microcurrent electrical stimulation (CES) vs sham CES over time on symptoms of depression, anxiety, fatigue, pain, and sleep disturbances in women with stage I-IIIA breast cancer receiving adjuvant chemotherapy.

Secondary

* To explore the relationships among selected markers of inflammation (e.g., tumor necrosis factor alpha, interleukin-6, interleukin-1β, and C-reactive protein), symptoms, and quality of life.
* To examine whether the symptoms of depression, anxiety, fatigue, sleep disturbances, and pain form a cluster.
* To examine the effects of CES on quality of life.

OUTLINE: Patients are stratified according to chemotherapy schedule (every 2 weeks for 8 courses vs every 3 weeks for 6 courses). Patients are randomized to 1 of 2 treatment arms.

* Arm I (cranial microcurrent electrical stimulation [CES]): Patients receive a CES unit (Alpha-Stim® 100 Microcurrent Stimulator) that passes microcurrent levels of biphasic electrical stimulation via ear-lobe electrodes. The CES unit is preset to provide 1 hour of 100 μA (sub-sensory level), modified square-wave biphasic stimulation on a 50% duty cycle at .05 Hz, and to automatically turn off at the end of 1 hour. Patients use their CES unit once daily in weeks 1-18.
* Arm II (sham CES): Patients receive a CES unit as in arm I, but the ear-lobe electrodes do not pass electrical current. Patients use their CES unit once daily in weeks 1-18.

Patients complete symptom questionnaires (e.g., the Hospital Anxiety and Depression Scale, the Brief Pain Inventory Short-Form, the Brief Fatigue Inventory, and the General Sleep Disturbance Scale) weekly in weeks 1-18. Patients also complete a quality-of-life questionnaire in weeks 1, 7, and 18.

Blood samples are collected in weeks 1, 7, and 18 and analyzed for cytokines (e.g., tumor necrosis factor alpha, interleukin-6, and interleukin-1β) and C-reactive protein.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of stage I-IIIA breast cancer
* Scheduled to receive adjuvant chemotherapy
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

* Pre, peri, or post-menopausal
* ECOG performance status 0-1
* No dementia
* No active psychosis
* No history of seizure disorder
* No implanted electrical device

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior chemotherapy
* No initiation of a medication regimen for depression or other psychiatric condition within the past 30 days

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2009-04; Primary Completion 2013-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deborah McGuire, PhD,RN,FAAN, Principal Investigator — Massey Cancer Center

REFERENCES:
- [Derived] Lyon D, Kelly D, Walter J, Bear H, Thacker L, Elswick RK. Randomized sham controlled trial of cranial microcurrent stimulation for symptoms of depression, anxiety, pain, fatigue and sleep disturbances in women receiving chemotherapy for early-stage breast cancer. Springerplus. 2015 Jul 23;4:369. doi: 10.1186/s40064-015-1151-z. eCollection 2015. PMID 26435889

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Women with stage I to IIIA breast cancer scheduled to receive chemotherapy with a performance score <2 recruited from five Cancer Centers across Virginia. Previous chemotherapy, dementia or active psychosis, seizure disorder, implanted electrical device, or taking medication psychiatric condition with 30 days prior to enrollment were excluded.
Pre-assignment Details: Following completion of informed consent study participants were stratified by initial chemotherapy regimen (dose dense versus non-dose dense) and then randomly assigned to one of two groups: actual or sham CES.
Period: Overall Study
Arm/Group | Arm I (Cranial Microcurrent Electrical Stimulation [CES]) | Arm II (Sham CES)
Started | 81 | 80
Completed | 77 | 75
Not Completed | 4 | 5
Not completed — Too overwhelmed by treatment | 2 | 5
Not completed — Adverse Event | 1 | 0
Not completed — No post baseline data | 1 | 0

BASELINE CHARACTERISTICS:
Population: Patients who completed trial
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Cranial Microcurrent Electrical Stimulation [CES]) | Arm II (Sham CES) | Total
Number analyzed (Participants) | 77 | 75 | 152
Age, Continuous [Median (Standard Deviation); unit: years] | 51.03 (11.06) | 51.41 (8.55) | 51.22 (9.805)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 77 | 75 | 152
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 28 | 22 | 50
  White | 46 | 49 | 95
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 4 | 7
Region of Enrollment [Number; unit: participants]
  United States | 77 | 75 | 152
Stage of Disease [Number; unit: participants] — Staged with TNM classifications. The TNM system is based on the size and/or extent (reach) of the primary tumor (T), the amount of spread to nearby lymph nodes (N), and the presence of metastasis (M) or secondary tumors formed by the spread of cancer cells to other parts of the body.
  participants
    Phase I | 16 | 18 | 34
    Phase II | 51 | 43 | 94
    Phase III | 10 | 14 | 24

OUTCOME MEASURES:

1. Primary Outcome: Effects of CES as Compared to Sham CES on Symptoms of Depression, Anxiety, Fatigue, Pain and Sleep Disturbances in Women Receiving Adjuvant Chemotherapy for Early-stage Breast Cancer
Description: Using Hospital Anxiety and Depression Scale (HADS) a 14 item scale, 7 relate to anxiety, 7 to depression; each item is scored from 0-3, a person can score 0 to 21 for either anxiety or depression (0 is best and 21 is worst), Brief Pain Inventory (BPI) short-form measures the intensity and interference of pain in the patient's life; 12 questions with 0 (does not interfere) to 10 (completely interferes); mean will be used as the measure of pain; Brief Fatigue Inventory (BFI) assess the severity and impact of cancer-related fatigue. Has 9 questions with 0 (does not interfere) to 10 (completely interferes), the total mean score is the mean of the 9 questions; severe fatigue can be defined as a score of 7 or higher, General Sleep Disturbance Scale (GSDS) 21 items to evaluate sleep issues (0=never to 7=every day); the 21 items are summed to produce a total score of 9=no sleep disturbance to 137=extreme sleep disturbance . Used standard questionnaire
Time Frame: Up to 2 weeks afer completion of study treatment, for up to 8 months
Measure: Least Squares Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm I (Cranial Microcurrent Electrical Stimulation [CES]) | Arm II (Sham CES)
Number analyzed (Participants) | 77 | 75
units on a scale
  Anxiety | 4.040 (0.419) | 4.529 (0.431)
  Depression | 4.520 (0.398) | 4.565 (0.407)
  Fatigue | 3.349 (0.294) | 3.191 (0.301)
  Pain | 1.174 (0.197) | 1.272 (0.202)
  Sleep | 38.235 (2.376) | 40.474 (2.443)

2. Secondary Outcome: To Examine Whether the Symptoms of Depression, Anxiety, Fatigue, Sleep Disturbances and Pain Form a Cluster.
Description: Examine correlations between the symptoms at baseline to determine a general pattern of association. Factor analysis (a statistical method used to describe variability among observed, correlated variables in terms of a potentially lower number of unobserved variables called factors) was performed to examine how these 5 symptoms cluster. A principal component factor analysis was performed on the correlation matrix for the symptom scores of anxiety, depression, pain, fatigue and sleep disturbance at up to two weeks after completion of study treatment, up to 8 months). For each analysis two factors were retained that explained 74% of the variability for the baseline symptom scores, 79% of the variability of the symptom scores at the midpoint and 78% of the variability in symptom scores at study completion. A varimax rotation was utilized and the factor loadings from the varimax rotation were reported.
Time Frame: up to 2 weeks after completion of study treatment, for up to 8 months
Measure: Number; unit: Rotated factor loading multiplied by 100
Groups:
- All Patients Analyzed: All patients
Arm/Group | All Patients Analyzed
Number analyzed (Participants) | 152
Rotated factor loading multiplied by 100
  Anxiety Factor 1 Loading-Baseline | 20
  Anxeity Factor 2 Loading-Baseline | 85
  Anxiety Factor 1 Loading-Midpoint Chemotherapy | 89
  Anxiety Factor 2 Loading-Midpoint Chemotherapy | 9
  Anxiety Factor 1 Loading-Post Chemotherapy | 88
  Anxiety Factor 2 Loading-Post Chemotherapy | 22
  Depression Factor 1 Loading-Baseline | 16
  Depression Factor 2 Loading-Baseline | 87
  Depression Factor 1 Loading-Midpoint Chemotherapy | 76
  Depression Factor 2 Loading-Midpoint Chemotherapy | 43
  Depression Factor 1 Loading-Post Chemotherapy | 86
  Depression Factor 2 Loading-Post Chemotherapy | 31
  Fatigue Factor 1 Loading-Baseline | 85
  Fatigue Factor 2 Loading-Baseline | 16
  Fatigue Factor 1 Loading-Midpoint Chemotherapy | 63
  Fatigue Factor 2 Loading-Midpoint Chemotherapy | 59
  Fatigue Factor 1 Loading-Post Chemotherapy | 44
  Fatigue Factor 2 Loading-Post Chemotherapy | 73
  Pain Factor 1 Loading-Baseline | 83
  Pain Factor 2 Loading-Baseline | 12
  Pain Factor 1 Loading-Midpoint Chemotherapy | 18
  Pain Factor 2 Loading-Midpoint Chemotherapy | 94
  Pain Factor 1 Loading-Post Chemotherapy | 13
  Pain Factor 2 Loading-Post Chemotherapy | 89
  Sleep Factor 1 Loading-Baseline | 67
  Sleep Factor 2 Loading-Baseline | 48
  Sleep Factor 1 Loading-Midpoint Chemotherapy | 79
  Sleep Factor 2 Loading-Midpoint Chemotherapy | 31
  Sleep Factor 1 Loading-Post Chemotherapy | 52
  Sleep Factor 2 Loading-Post Chemotherapy | 67

3. Secondary Outcome: Means and Standard Deviations of Biomarkers Log(CRP pg/ml), Log(IL-1b pg/ml), Log(IL-6 pg/ml) and Log(TNF-a pg/ml).
Description: Simple correlations will be computed at Midpoint Chemotherapy for the log transformed biomarker values; IL1-β, IL-6, TNF-α, CRP. These are the biomarkers of inflammation.
Time Frame: Baseline
Population: Per protocol, for all subjects with available data. No imputation was utilized.
Measure: Mean (Standard Deviation); unit: Log(pg/ml)
Groups:
- Arm I: Cranial Microcurrent Electrical Stimulation (CES)
- Arm II: Sham CES
Arm/Group | Arm I | Arm II
Number analyzed (Participants) | 77 | 75
Log(pg/ml)
  Log(CRP pg/ml) | 28.64 (1.67) | 28.92 (1.32)
  Log(IL-1b pg/ml) | 9.88 (69.85) | 32.60 (259.03)
  Log(IL-6 pg/ml) | 0.33 (2.65) | 0.09 (3.21)
  Log(TNF-a pg/ml) | -0.63 (3.49) | -0.19 (3.49)
Statistical Analysis 1: Comparison: Arm I vs Arm II; Spearman correlation coefficients were computed for the biomarkers. P-Values shown are not adjusted for multiple comparisons. The a priori threshold for statistical significance was P less than 0.05. This information applies to all rows listed in the table; Test type: Superiority or Other; p < 0.05, t-test, 2 sided

4. Secondary Outcome: Relationships Among Biomarkers Log(CRP pg/ml), Log(IL-1b pg/ml), Log(IL-6 pg/ml) and Log(TNF-a pg/ml).
Description: Simple correlations will be computed at Baseline for the log transformed biomarker values; IL1-β, IL-6, TNF-α, CRP. These are the biomarkers of inflammation.
Time Frame: Baseline
Measure: Number; unit: correlation coefficient
Arm/Group | All Patients Analyzed
Number analyzed (Participants) | 152
correlation coefficient
  Correlation between Log (CRP)-Log (IL-1B) | 0.031
  Correlation between Log (CRP)-Log IL6) | 0.243
  Correlation between Log (CRP)-Log (TNF-a) | 0.002
  Correlation between Log (IL-1B)-Log (IL6) | 0.453
  Correlation between Log (IL-1B)-Log (TNF-a) | 0.570
  Correlation between Log (IL6)-Log (TNF-a) | 0.320

5. Secondary Outcome: Relationships Among Anxiety, Depression, Fatigue, Pain and Sleep Scores - Means at Baseline
Description: Measured using Hospital Anxiety and Depression Scale (HADS) a fourteen item scale, 7 relate to anxiety and 7 to depression; each item is scored from 0-3, this means a person can score 0 to 21 for either anxiety or depression (0 is best and 21 is worst), Brief Pain Inventory (BPI) short-form measures the intensity of pain and interference of pain in the patient's life; 12 questions with 0 (does not interfere) to 10 (completely interferes); mean will be used as the measure of pain; Brief Fatigue Inventory (BFI) assess the severity and impact of cancer-related fatigue. it has 9 questions with 0 (does not interfere) to 10 (completely interferes); severe fatigue can be defined as a score of 7 or higher, General Sleep Disturbance Scale (GSDS) 21 items to evaluate sleep issues (0=never to 7=every day); the 21 items are summed to produce a total score of 9=no sleep disturbance to 137=extreme sleep disturbance . Used standard questionnaire scoring system.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm I | Arm II
Number analyzed (Participants) | 77 | 75
units on a scale
  Anxiety | 7.09 (4.09) | 7.59 (4.13)
  Depression | 3.03 (2.48) | 3.06 (2.78)
  Fatigue | 1.95 (2.71) | 2.63 (2.89)
  Pain | 1.24 (2.05) | 1.45 (1.98)
  Sleep | 40.70 (24.83) | 40.30 (23.87)

6. Secondary Outcome: Relationships Among Symptom Scores - Correlations at Baseline Chemotherapy
Description: Simple correlations will be computed at Baseline Chemotherapy for symptoms.
Time Frame: Baseline
Measure: Number; unit: correlation coefficient
Arm/Group | All Patients Analyzed
Number analyzed (Participants) | 152
correlation coefficient
  Correlation between Anxiety-Depression | 0.610
  Correlation between Anxiety-Fatigue | 0.303
  Correlation between Anxiety-Pain | 0.298
  Correlation between Anxiety-Sleep | 0.474
  Correlation between Depression-Fatigue | 0.343
  Correlation between Depression-Pain | 0.315
  Correlation between Depression-Sleep | 0.488
  Correlation between Fatigue-Pain | 0.482
  Correlation between Fatigue-Sleep | 0.492
  Correlation between Pain-Sleep | 0.388

7. Secondary Outcome: Relationships Among Quality of Life Scores - Means at Baseline
Description: Measured using the Functional Assessment of Cancer Therapy for Patients with Breast Cancer (FACT-B). A 44-item self-report instrument designed to measure multidimensional quality of life in patient with breast cancer. 0=not at all to 4=very much. Utilized standard questionnaire scoring system. The items are summed to produce a total score 0=not at all to 176=very much. The FACT-B BCA has 10 questions that range from 0 (not at all) to 4 (very much); thus the FACT-B BCA ranges from 0 to 40. Both the FACT-B and FACT-BCA are scored so that high scores indicate higher levels of quality of life.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm I | Arm II
Number analyzed (Participants) | 77 | 75
units on a scale
  FACT-B Total | 113.44 (17.65) | 111.83 (17.91)
  FACT-B BCA Specific | 27.42 (5.05) | 26.05 (6.04)

8. Secondary Outcome: Relationships Among Quality of Life Scores - Correlations at Baseline
Description: Simple correlations will be computed at Baseline for quality of life scores.
Time Frame: Baseline
Measure: Number; unit: correlation coefficient
Arm/Group | All Patients Analyzed
Number analyzed (Participants) | 152
correlation coefficient | 0.744

9. Secondary Outcome: Mean and Standard Deviation of Biomarkers Log(CRP pg/ml), Log(IL-1b pg/ml), Log(IL-6 pg/ml) and Log(TNF-a pg/ml).
Description: as for outcome 3
Time Frame: Midpoint Chemotherapy, up to 4 months
Measure: Mean (Standard Deviation); unit: Log (pg/ml)
Arm/Group | Arm I | Arm II
Number analyzed (Participants) | 77 | 75
Log (pg/ml)
  Log (CRP) | 28.62 (1.69) | 29.09 (1.18)
  Log (IL-1B) | 6.52 (52.59) | 24.68 (171.81)
  Log (IL6) | -0.22 (2.91) | 0.55 (2.80)
  Log (TNF-a) | -0.89 (3.52) | -0.15 (3.68)

10. Secondary Outcome: Relationships Among Biomarkers Log (CRP), Log (IL-1B), Log (IL6), and Log (TNF-a) - Correlations at Midpoint Chemotherapy
Description: as for outcome 3
Time Frame: Midpoint Chemotherapy, up to 4 months
Measure: Number; unit: correlation coefficient
Arm/Group | All Patients Analyzed
Number analyzed (Participants) | 152
correlation coefficient
  Correlation between Log (CRP)-Log (IL-1B) | 0.060
  Correlation between Log (CRP)-Log IL6) | 0.337
  Correlation between Log (CRP)-Log (TNF-a) | 0.102
  Correlation between Log (IL-1B)-Log (IL6) | 0.390
  Correlation between Log (IL-1B)-Log (TNF-a) | 0.593
  Correlation between Log (IL6)-Log (TNF-a) | 0.298

11. Secondary Outcome: Relationships Among Anxiety, Depression, Fatigue, Pain and Sleep Scores - Means at Midpoint Chemotherapy
Description: as for outcome 5
Time Frame: Midpoint Chemotherapy, up to 4 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm I | Arm II
Number analyzed (Participants) | 77 | 75
units on a scale
  Anxiety | 4.40 (3.19) | 4.98 (3.72)
  Depression | 4.24 (3.22) | 4.02 (3.14)
  Fatigue | 3.15 (2.21) | 3.14 (2.39)
  Pain | 1.25 (1.44) | 1.09 (1.56)
  Sleep | 38.70 (18.28) | 42.44 (21.73)

12. Secondary Outcome: Relationships Among Symptom Scores - Correlations at Midpoint Chemotherapy
Description: Simple correlations will be computed at Midpoint Chemotherapy for symptoms.
Time Frame: Midpoint Chemotherapy, up to 4 months
Measure: Number; unit: correlation coefficient
Arm/Group | All Patients Analyzed
Number analyzed (Participants) | 152
correlation coefficient
  Correlation between Anxiety-Depression | 0.723
  Correlation between Anxiety-Fatigue | 0.512
  Correlation between Anxiety-Pain | 0.305
  Correlation between Anxiety-Sleep | 0.604
  Correlation between Depression-Fatigue | 0.632
  Correlation between Depression-Pain | 0.412
  Correlation between Depression-Sleep | 0.624
  Correlation between Fatigue-Pain | 0.507
  Correlation between Fatigue-Sleep | 0.719
  Correlation between Pain-Sleep | 0.429

13. Secondary Outcome: Relationships Among Quality of Life Scores - Means at Midpoint Chemotherapy
Description: as for outcome 7
Time Frame: Midpoint Chemotherapy, up to 4 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm I | Arm II
Number analyzed (Participants) | 77 | 75
units on a scale
  FACT-B Total | 111.57 (18.35) | 108.45 (22.46)
  FACT-B BCA Specific | 26.96 (5.47) | 25.96 (5.39)

14. Secondary Outcome: Relationships Among Quality of Life Scores - Correlations at Midpoint Chemotherapy
Description: Simple correlations will be computed at Midpoint Chemotherapy for quality of life scores.
Time Frame: Midpoint Chemotherapy, up to 4 months
Measure: Number; unit: correlation coefficient
Arm/Group | All Patients Analyzed
Number analyzed (Participants) | 152
correlation coefficient | 0.743

15. Secondary Outcome: Mean and Standard Deviation of Biomarkers Log(CRP pg/ml), Log(IL-1b pg/ml), Log(IL-6 pg/ml) and Log(TNF-a pg/ml).
Description: Simple correlations will be computed after completion of study treatment for the log transformed biomarker values; IL1-β, IL-6, TNF-α, CRP. These are the biomarkers of inflammation.
Time Frame: Up to 2 weeks after completion of study treatment, for up to 8 months
Measure: Mean (Standard Deviation); unit: Log (pg/ml)
Arm/Group | Arm I | Arm II
Number analyzed (Participants) | 77 | 75
Log (pg/ml)
  Log (CRP) | 28.64 (1.26) | 29.00 (1.32)
  Log (IL-1B) | 10.50 (83.81) | 1.35 (5.65)
  Log (IL6) | 0.68 (2.29) | 0.73 (2.26)
  Log (TNF-a) | -1.34 (3.64) | -0.33 (3.22)

16. Secondary Outcome: Relationships Among Biomarkers Log (CRP), Log (IL-1B), Log (IL6), and Log (TNF-a) - Correlations at End of Treatment
Description: Simple correlations will be computed at Chemotherapy End of Treatment for the log transformed biomarker values; IL1-β, IL-6, TNF-α, CRP. These are the biomarkers of inflammation.
Time Frame: Up to 2 weeks afer completion of study treatment, for up to 8 months
Measure: Number; unit: correlation coefficient
Arm/Group | All Patients Analyzed
Number analyzed (Participants) | 152
correlation coefficient
  Correlation between Log (CRP)-Log (IL-1B) | 0.057
  Correlation between Log (CRP)-Log IL6) | 0.343
  Correlation between Log (CRP)-Log (TNF-a) | 0.135
  Correlation between Log (IL-1B)-Log (IL6) | 0.383
  Correlation between Log (IL-1B)-Log (TNF-a) | 0.464
  Correlation between Log (IL6)-Log (TNF-a) | 0.134

17. Secondary Outcome: Relationships Among Anxiety, Depression, Fatigue, Pain and Sleep Scores - Means at End of Chemotherapy
Description: as for outcome 5
Time Frame: Up to 2 weeks afer completion of study treatment, for up to 8 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm I | Arm II
Number analyzed (Participants) | 77 | 75
units on a scale
  Anxiety | 4.07 (3.51) | 4.51 (4.04)
  Depression | 4.47 (3.36) | 4.63 (3.67)
  Fatigue | 3.34 (2.47) | 3.32 (2.55)
  Pain | 1.14 (1.65) | 1.32 (1.80)
  Sleep | 38.50 (20.19) | 40.91 (21.21)

18. Secondary Outcome: Relationships Among Symptom Scores - Correlations at End of Chemotherapy
Description: Simple correlations will be computed at end of Chemotherapy for symptoms.
Time Frame: Up to 2 weeks afer completion of study treatment, for up to 8 months
Measure: Number; unit: correlation coefficient
Arm/Group | All Patients Analyzed
Number analyzed (Participants) | 152
correlation coefficient
  Correlation between Anxiety-Depression | 0.678
  Correlation between Anxiety-Fatigue | 0.467
  Correlation between Anxiety-Pain | 0.409
  Correlation between Anxiety-Sleep | 0.515
  Correlation between Depression-Fatigue | 0.564
  Correlation between Depression-Pain | 0.368
  Correlation between Depression-Sleep | 0.637
  Correlation between Fatigue-Pain | 0.488
  Correlation between Fatigue-Sleep | 0.643
  Correlation between Pain-Sleep | 0.484

19. Secondary Outcome: Effects of Treatment on Quality of Life - Means at End of Treatment
Description: Measured using the Functional Assessment of Cancer Therapy for Patients with Breast Cancer (FACT-B). A 44-item self-report instrument designed to measure multidimensional quality of life in patient with breast cancer. 0=not at all to 4=very much. Utilized standard questionnaire scoring system. The items are summed to produce a total score 0=not al all to 176=very much. The FACT-B BCA has 10 questions that range from 0 (not at all) to 4 (very much); thus the FACT-B BCA ranges from 0 to 40. Both the FACT-B and FACT-BCA are scored so that high scores indicate higher levels of quality of life.
Time Frame: up to 2 weeks after completion of study treatment, for up to 8 months
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Arm I (Cranial Microcurrent Electrical Stimulation [CES]) | Arm II (Sham CES)
Number analyzed (Participants) | 77 | 75
units on a scale
  Total Score | 108.11 (2.52) | 105.96 (2.59)
  Breast Cancer Specific | 25.51 (0.75) | 24.66 (0.77)

20. Secondary Outcome: Relationships Among Quality of Life Scores - Correlations at End of Chemotherapy
Description: Simple correlations will be computed at End of Chemotherapy for quality of life scores.
Time Frame: Up to 2 weeks afer completion of study treatment, for up to 8 months
Measure: Number; unit: correlation coefficient
Arm/Group | All Patients Analyzed
Number analyzed (Participants) | 152
correlation coefficient | 0.772

ADVERSE EVENTS:
Time Frame: Up to 20 weeks
Arm/Group | Arm I (Cranial Microcurrent Electrical Stimulation [CES]) | Arm II (Sham CES)
Serious Adverse Events (participants affected / at risk) | 1/77 | 0/75
Other Adverse Events (participants affected / at risk) | 0/77 | 0/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Cranial Microcurrent Electrical Stimulation [CES]) (N=77) | Arm II (Sham CES) (N=75)
Seizure (Nervous system disorders) | 1 (1) | 0 (0) — nonstudy related

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No